CLINICAL TRIAL: NCT05642299
Title: Multimodal EEG and NIRS-based BCI With Assistive Soft Robotics for Stroke
Brief Title: Multimodal EEG and NIRS-based BCI With Assistive Soft Robotics for Stroke (MBCI-SR)
Acronym: MBCI-SR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Institute for Infocomm Research (Other); Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Chloe Chung Lau Ha, Principal Physiotherapist, Tan Tock Seng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/00715
Record Dates: First submitted 2022-11-15; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Stroke
Keywords: Brain-Computer Interface; upper limb rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBCI-SR (Experimental): BCI based robotic rehabilitation works by detecting the motor intent of the user from Electroencephalogram signals to drive rehabilitation assisted by the soft robotics gloves.
  Interventions: Device: MBCI-SR

INTERVENTIONS:
Device: MBCI-SR — Participants will be asked to wear and EEG+NIRS cap and a soft robotic glove on their stroke-impaired hand. The participant will be instructed to ask to imagine to picture moving the stroke-imparied hand in the mind. The brain signal (EEG and NIRS data) will be recorded as a reference. When the participant pictures this move again, upon detection of such imagined move by MBCI-SR system, the glove will be activated and assists the participants to perform a specific upper limb task based on individual ability. There are six different activities of daily living (ADL)-oriented tasks enacted through a virtual arm and virtual objects, which formed the visual feedback for the participants. These tasks include scanning goods, moving an object upward to a cabinet, using two hands to move a towel, pouring of water into a cup, eating action and fine motor movement of picking up a small block using two fingers. Training intensity is 1.5 hours for 3 times a week for 6 weeks, a total of 18 sessions.

SUMMARY:
One-third of patients who had stroke suffered persistent disabilities, and upper limb (UL) motor impairment is one of the main disabilities. Recent clinical studies had been conducted using non-invasive EEG-based BCI via motor imagery, for post-stroke rehabilitation, yielded motor improvement of 7.2 on the Fugl-Meyer Motor Assessment (FMA-UE)score in chronic stroke patients that is significantly better than standard care. However, all the stroke patients underwent the same "one-size-fits-all" treatment option involving all six different activities of daily living (ADL)-oriented tasks regardless of their impairment or ability.

Investigators hypothesize that precision personalized stroke rehabilitation intervention that is tailored to the patient hold more promise than a "one-size-fits-all" stroke rehabilitation strategy.

DETAILED DESCRIPTION:
1. To address the "one-size-fits-all" stroke rehabilitation strategy, RRIS will develop an Ability data-driven personalized stroke rehabilitation based on the stroke patient's UL impairment and motor ability, by first matching 6 UL tasks in RRIS Ability Database with the 6 ADL tasks of the BCI-SR Intervention via similarity indices. A personalized subset of ADL tasks treatment options is then generated by a data-driven recommendation based on the patient's ability, movement pattern of the treatment option and the normative data from the RRIS Ability Database. A multi-modal BCI is proposed to perform EEG subject-specific calibration using Near-infrared spectroscopy, NIRS to ensure motor imagery compliance.
2. stroke subjects with UL impairments (score 11-45 on the FMA-UE) will be recruited to undergo the UL tasks assessment at RRIS. They will then undergo the personalized stroke rehabilitation using the Multimodal EEG and NIRS-based BCI with Soft Robotic therapy for 1.5 hour over 6 weeks, 3 times a week. The effectiveness of the personalized stroke rehabilitation can then be retrospectively compared to the use of "one-size-fits-all" ADL tasks in the previous clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* first ever stroke prior to clinical trial
* Fugl-Meyer Assessment scale of upper extremity impairment of 11-45 out of a maximum score of 66
* ability to give own consent
* ability to pay attention and maintain supported sitting for 1.5 hours continuously
* able to comprehend and follow commands
* fulfils BCI resting brain states on initial screening
* unilateral upper limb impairment

Exclusion Criteria:

* recurrent stroke
* inability to follow command and sit upright for 1.5 hours
* hemi-spatial neglect
* spasticity assessed by Modified Ashworth Scale more than 2/4
* History of Epilepsy
* Fixed contracture / deformity of finger joints
* upper limb pain impeding movements with visual analogy scale > 4/10
* Severe aphasia or cognitive impairment despite visual aids
* other conditions ensuing upper limb weakness
* poor skin conditions
* skull defect that might affect EEG or NIRS reading
* allergy to electrodes or adhesive gel
* significant vision and hearing impairment affecting participation
* Pregnant women

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-09-14 (Estimated); Study Completion 2023-12-14 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer score of upper limb | Baseline
  a measure for upper extremity, movement coordination and reflex action.
Fugl-Meyer score of upper limb | at week 4 (mid point)
  a measure for upper extremity, movement coordination and reflex action.
Fugl-Meyer score of upper limb | at week 6 (completion of intervention)
  a measure for upper extremity, movement coordination and reflex action.
Fugl-Meyer score of upper limb | at week 12 (at 3 month post intervention)
  a measure for upper extremity, movement coordination and reflex action.
Fugl-Meyer score of upper limb | at week 24 (at 6 month post intervention)
  a measure for upper extremity, movement coordination and reflex action.

SECONDARY OUTCOMES:
Action Research Arm Test | Baseline
  A measure for upper extremity functioning, such as dexterity and motor coordination, the key components in performing ADLs
Action Research Arm Test | at week 12 (at 3 months post intervention)
  A measure for upper extremity functioning, such as dexterity and motor coordination, the key components in performing ADLs
Action Research Arm Test | at week 24 ( at 6 months post intervention)
  A measure for upper extremity functioning, such as dexterity and motor coordination, the key components in performing ADLs

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Lauha Chung, PhD, Principal Investigator — Tan Tock Seng Hospital; Kai Keng Ang, Principal Investigator — Institute for Infocomm Research
Locations (1):
- Tan Tock Seng Hospital Rehabilitation Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Share the study protocol, clinical study report and results

REFERENCES:
- [Background] Daly JJ, Wolpaw JR. Brain-computer interfaces in neurological rehabilitation. Lancet Neurol. 2008 Nov;7(11):1032-43. doi: 10.1016/S1474-4422(08)70223-0. Epub 2008 Oct 2. PMID 18835541
- [Result] Ang KK, Chua KS, Phua KS, Wang C, Chin ZY, Kuah CW, Low W, Guan C. A Randomized Controlled Trial of EEG-Based Motor Imagery Brain-Computer Interface Robotic Rehabilitation for Stroke. Clin EEG Neurosci. 2015 Oct;46(4):310-20. doi: 10.1177/1550059414522229. Epub 2014 Apr 21. PMID 24756025
- [Result] Ang KK, Guan C, Phua KS, Wang C, Zhou L, Tang KY, Ephraim Joseph GJ, Kuah CW, Chua KS. Brain-computer interface-based robotic end effector system for wrist and hand rehabilitation: results of a three-armed randomized controlled trial for chronic stroke. Front Neuroeng. 2014 Jul 29;7:30. doi: 10.3389/fneng.2014.00030. eCollection 2014. PMID 25120465
- [Result] Cheng N, Phua KS, Lai HS, Tam PK, Tang KY, Cheng KK, Yeow RC, Ang KK, Guan C, Lim JH. Brain-Computer Interface-Based Soft Robotic Glove Rehabilitation for Stroke. IEEE Trans Biomed Eng. 2020 Dec;67(12):3339-3351. doi: 10.1109/TBME.2020.2984003. Epub 2020 Nov 19. PMID 32248089
- [Result] Ang KK, Guan C, Chua KS, Ang BT, Kuah CW, Wang C, Phua KS, Chin ZY, Zhang H. A large clinical study on the ability of stroke patients to use an EEG-based motor imagery brain-computer interface. Clin EEG Neurosci. 2011 Oct;42(4):253-8. doi: 10.1177/155005941104200411. PMID 22208123